CLINICAL TRIAL: NCT04988165
Title: Clinical Study on Prevention and Treatment of Pyrotinib Associated Diarrhea With Traditional Chinese Medicine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCM-padia001
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Diarrhea Caused by Antitumor Drugs
Keywords: Diarrhea; Pyrotinib; Traditional Chinese Medicine
MeSH Terms: conditions — Diarrhea | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Traditional Chinese Medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — It is a common prescription used in traditional Chinese medicine to treat diarrhea with remarkable efficacy.

SUMMARY:
Pyrotinib is an important drug for the treatment of breast cancer, but the incidence of diarrhea is very high. At present, there is no particularly effective drug for diarrhea induced by pyrotinib. Trying to intervene with traditional Chinese medicine may bring better results to patients.

DETAILED DESCRIPTION:
Pyrotinib is an important drug for the treatment of breast cancer, but the incidence of diarrhea is very high. At present, there is no particularly effective drug for diarrhea induced by pyrotinib. Trying to intervene with traditional Chinese medicine may bring better results to patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet the following two conditions:

  1. Planned administration of pyrotinib ≥ 21 days;
  2. Grade 1-3 diarrhea after taking pyrotinib, and it is planned to continue taking pyrotinib;

     2. Age ≥ 18 years old;

     3. ECOG PS 0-2；

     4. Life expectancy ≥ 6 months;

     5. Voluntarily join the study, sign informed consent, have good compliance and are willing to cooperate with follow-up

     Exclusion Criteria:

  <!-- -->

  1. Those who may be allergic to pyrotinib or excipients;
  2. It has many factors affecting the absorption of oral drugs, such as inability to swallow, nausea and vomiting, etc;
  3. Patients with biliary obstruction;
  4. Participate in other diarrhea related clinical trials;
  5. Female patients during pregnancy and lactation, female patients with fertility and positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptives during the whole test period;
  6. according to the researchers' judgment, there are serious diseases that endanger the safety of patients, or affect the patients to complete the study (including, but not limited to, severe hypertension and severe diabetes, which can not be controlled by drugs).
  7. Any other circumstances in which the investigator believes that the patient is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2022-10-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
incidence of grade 3-4 diarrhea | From the beginning of taking traditional Chinese medicine to the 21st day
  The number of stools per day increased by ≥ 7 compared with baseline; Incontinence, indication of hospitalization; Compared with baseline, the yield of stoma increased significantly; Daily activities are limited.Life threatening diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: zhongsheng tong, doctor, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD is under construction